CLINICAL TRIAL: NCT05935384
Title: SIBYL: obServation of Therapy Response With lIquid BiopsY evaLuation
Status: Recruiting | Type: Observational
Sponsor: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-MX-001
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Non-small Cell Lung Cancer; Colorectal Cancer; Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Cohort 1: Unresectable Stage III/IV NSCLC: Blood samples collected will be banked
  Interventions: Diagnostic Test: Guardant360
- Cohort 2: Stage IV Colorectal: Blood samples collected will be banked
  Interventions: Diagnostic Test: Guardant360
- Cohort 3: Unresectable Stage III/IV Breast - HR+ HER2-: Blood samples collected will be banked
  Interventions: Diagnostic Test: Guardant360
- Cohort 4: Unresectable Stage III/IV Breast - HR- HER2+: Blood samples collected will be banked
  Interventions: Diagnostic Test: Guardant360
- Cohort 5: Unresectable Stage III/IV Breast - HR+ HER2+: Blood samples collected will be banked
  Interventions: Diagnostic Test: Guardant360
- Cohort 6: Unresectable Stage III/IV Breast - Triple Negative: Blood samples collected will be banked
  Interventions: Diagnostic Test: Guardant360

INTERVENTIONS:
Diagnostic Test: Guardant360 — Guardant360 is a qualitative next generation sequencing (NGS)-based in vitro diagnostic device for detection of single nucleotide variants (SNVs), insertions and deletions (indels), copy number amplifications (CNAs), and fusions in genes frequently mutated in cancer, using circulating cell-free DNA (cfDNA) obtained from the plasma of peripheral whole blood collected in Streck Cell-Free DNA Blood Collection Tubes.

SUMMARY:
The purpose of SIBYL is to generate clinical validity data for the ability of a future version of Guardant360 developed by Guardant Health to measure response to systemic therapy in patients with unresectable advanced solid tumors. It is necessary to collect clinical data points and treatment outcomes in order to demonstrate clinical validity for longitudinal monitoring with ctDNA and correlation of ctDNA dynamics with therapeutic response, as evaluated by standard methods, including RECIST 1.1 and CT scan measurements.

ELIGIBILITY:
Inclusion Criteria

Each participant must satisfy all the following criteria to be enrolled in the study:

1. Age ≥18 years old
2. Are treated with systemic therapy and/or oral SOC regimen at the site of enrollment during entirety of study
3. Patient is either treatment naive and has not yet commenced first line SOC therapy OR patient has completed first line SOC therapy and will commence second line of SOC therapy
4. Able to understand, and capable of providing written consent to participate in the study
5. Are willing to have de-identified clinical data shared with investigators at regular intervals outlined in the study protocol and informed consent
6. Are willing to provide blood samples at enrollment and at subsequent clinical visits
7. Have a histologically confirmed Index cancer that qualifies for inclusion, defined as:

   * Cohort 1: Unresectable Stage III/IV NSCLC (~125)
   * Cohort 2: Stage IV Colorectal (~125)
   * Cohort 3: Unresectable Stage III/IV Breast - HR+ HER2- (~55)
   * Cohort 4: Unresectable Stage III/IV Breast - HR- HER2+ (~55)
   * Cohort 5: Unresectable Stage III/IV Breast - HR+ HER2+ (~55)
   * Cohort 6: Unresectable Stage III/IV Breast - Triple Negative (~55) Determination of stage for eligibility assessment and enrollment should be based on clinical or pathologic stage.

Exclusion Criteria

Any potential participant who meets and of the following criteria at the time of initial enrollment will be excluded from participating in the study:

1. History of prior solid malignancy or hematological malignancy within five years of enrollment
2. Life expectancy ≤12 weeks
3. Unable to collect a baseline blood sample during a SOC venipuncture, and prior to starting SOC regimen
4. Is participating in a clinical trial or another observational study that is evaluating the performance of another genomic test for detecting/predicting clinical response/progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary study population will include participants with Non-small cell lung cancer (stage III-IV), Colorectal adenocarcinoma (stage III-IV), and Breast Cancer (stage III-IV), as per inclusion/exclusion criteria. Approximately 470 total patients will be enrolled into the study.
Sampling Method: Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of ctDNA to Detect Disease Progression | 6 years
  The Primary Endpoint, sensitivity of ctDNA to detect disease progression, will be evaluated from all eligible subjects within the primary study cohorts (breast cancer, NSCLC, or CRC)

SECONDARY OUTCOMES:
RECIST Response | 6 years
  RECIST v1.1 response: defined as the tumor response to treatment as measured by restaging scans in subjects who have increasing or decreasing ctDNA quantities before the time of scan and correlating this change with the clinical response
Progression-Free Survival (PFS) | 6 years
  PFS: defined as the quantitative changes in ctDNA that correlate or associate with participant's progression free survival on each line of SOC therapy
Lead Time | 6 years
  Lead time: defined as the interval between ctDNA detection or increase and clinical detection of disease progression

CONTACTS AND LOCATIONS:
Locations (1):
- Orchard Healthcare Research Inc., Skokie, Illinois, United States

IPD SHARING:
Plan to Share IPD: No